CLINICAL TRIAL: NCT06920485
Title: Clinical and Microbiological Evaluation of the Effects of Hypochlorous Acid Mouthwash Use in the Postoperative Period of Mandibular Third Molar Tooth Extractions
Brief Title: Effect of Hypochlorous Acid-containing Mouthwash on Healing After Impacted Wisdom Tooth Surgery
Acronym: Mouthwash
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Özgün Yıldırım, Doctor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06.02.2025-2025/3-25/1
Record Dates: First submitted 2025-03-19; First posted 2025-04-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Oral Health
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hypochlorous acid (Experimental): Wound healing and microbiological analysis will be performed by administering hypochlorous acid to this group.
  All surgical procedures will be performed under local anesthesia (80 mg articaine hydrochloride and 0.02 mg epinephrine, Maxicaine Fort ampoule, Vem İlaç, İstanbul, Turkey) and sterile conditions following the application of inferior alveolar block anesthesia + buccal mucosa anesthesia. Osteotomy (bone removal) and, if necessary, root dissection will be performed using a surgical handpiece with sterile saline solution and irrigation. Following tooth extraction, the socket will be checked and any sharp bone protrusions will be removed. The area will be closed primarily using non-resorbable silk suture material (surgical silk suture, 3/0, Doğsan, Turkey).
  Interventions: Procedure: Third molar surgery; Diagnostic Test: Pain Medicine; Diagnostic Test: Wound healing; Other: Total bacterial load
- Chlorhexidine gluconate (Experimental): Wound healing and microbiological analysis will be performed by administering chlorhexidine gluconate to this group.
  All surgical procedures will be performed under local anesthesia (80 mg articaine hydrochloride and 0.02 mg epinephrine, Maxicaine Fort ampoule, Vem İlaç, İstanbul, Turkey) and sterile conditions following the application of inferior alveolar block anesthesia + buccal mucosa anesthesia. Osteotomy (bone removal) and, if necessary, root dissection will be performed using a surgical handpiece with sterile saline solution and irrigation. Following tooth extraction, the socket will be checked and any sharp bone protrusions will be removed. The area will be closed primarily using non-resorbable silk suture material (surgical silk suture, 3/0, Doğsan, Turkey).
  Interventions: Procedure: Third molar surgery; Diagnostic Test: Pain Medicine; Diagnostic Test: Wound healing; Other: Total bacterial load
- Physiological serum (Experimental): Wound healing and microbiological analysis will be performed by administering physiological serum to this group.
  All surgical procedures will be performed under local anesthesia (80 mg articaine hydrochloride and 0.02 mg epinephrine, Maxicaine Fort ampoule, Vem İlaç, İstanbul, Turkey) and sterile conditions following the application of inferior alveolar block anesthesia + buccal mucosa anesthesia. Osteotomy (bone removal) and, if necessary, root dissection will be performed using a surgical handpiece with sterile saline solution and irrigation. Following tooth extraction, the socket will be checked and any sharp bone protrusions will be removed. The area will be closed primarily using non-resorbable silk suture material (surgical silk suture, 3/0, Doğsan, Turkey).
  Interventions: Procedure: Third molar surgery; Diagnostic Test: Pain Medicine; Diagnostic Test: Wound healing; Other: Total bacterial load

INTERVENTIONS:
Procedure: Third molar surgery — Effects of different gargles/mouth rinses/antiseptic agents applied after impacted surgical tooth extraction on postoperative wound healing and total bacterial load
Diagnostic Test: Pain Medicine — After the extraction, patients will be given two separate forms with VAS scales for pain to mark every day for 7 days. The patient will be asked to mark the level of pain they feel on the scale. The amount of analgesic use on the home assessment form will also be recorded as part of the pain assessment. On the 7th day, healing in the wound area will also be assessed.
Diagnostic Test: Wound healing — The degree of healing of the wound area will be checked using Landry scoring.
Other: Total bacterial load — Total bacterial load will be evaluated by microbiological analysis of sutures obtained from all groups.

SUMMARY:
INTRODUCTION: Local chemotherapeutic agents are used to reduce inflammation after impacted tooth extraction and to minimize possible complications, as well as to increase patient comfort. The aim of this study is to compare the clinical and microbiological effects of different mouthwashes/mouth rinses/antiseptic agents applied after impacted surgical tooth extraction in patients with impacted mandibular third molars within the scope of pain, wound healing and total bacterial load criteria; postoperative complications and healing process.

MATERIAL AND METHODS: According to the Pell and Gregory classification, 96 volunteer patients with unilateral or bilateral Class 2 position A and B impacted mandibular third molars, being systemically healthy (ASA class 1), being between the ages of 18-45/young adult will participate in the study. The patients will be divided into 3 groups: Group 1, Patients who will be administered hypochlorous acid-containing mouthwash in addition to standard treatment after mandibular third molar surgery; Group 2, Patients who will be administered chlorhexidine gluconate-containing mouthwash in addition to standard treatment after mandibular third molar surgery; Group 3, Patients who will be administered sterile saline-containing mouthwash in addition to standard treatment after mandibular third molar surgery. Demographic data before the surgical procedure will be recorded in the patient follow-up form (Appendix-1). As a standard postoperative approach, all patients will be prescribed antibiotics (875 mg Amoxicillin+125 mg clavulonic acid, Augmentin-BID film-coated tablets, GlaxoSmithKline, Istanbul, Turkey), analgesics for use after surgery, and mouthwashes will be given depending on the groups. Patients will be asked to take antibiotics in the morning and evening for 5 days, use mouthwash for 7 days starting from the day after the procedure, and use mouthwash only when deemed necessary, and will be asked to record the amount they use on the home assessment form (ANNEX-2). All patients will be evaluated on the 7th day after the operation, and suture samples will be taken for microbiological load determination. All evaluations will be made before the operation and on the 7th day after the operation; and will be recorded on the patient assessment form (ANNEX-1). First of all, demographic information including age, gender, education level and the operation area will be recorded for all patients. Two separate forms with VAS scales for pain will be given to patients to mark every day for 7 days after the extraction. The patient will be asked to mark the level of pain they feel on the scale. The amount of analgesic use in the home assessment form will also be recorded within the scope of the pain assessment. Healing in the wound area will also be evaluated on the 7th day.

ELIGIBILITY:
Inclusion Criteria:

* Having a mandibular third molar with a unilateral or bilateral Class 2, Position A or B impaction according to the Pell and Gregory classification
* Being systemically healthy (ASA Class I)
* Aged between 18 and 45 years (young adult age group)
* Willingness to participate in the study

Exclusion Criteria:

* Age outside the specified range
* Pregnancy
* Currently breastfeeding
* Presence of infection in the third molar region (e.g., acute pericoronitis)
* Presence of cystic or tumoral lesions associated with the impacted third molar
* History of allergic reactions
* Presence of any systemic disease
* Unwillingness to participate in the study
* Poor oral hygiene that may negatively affect healing
* Smoking or alcohol addiction
* Use of antibiotics or mouthwash in the last three months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain levels after mandibular third molar surgery | From postoperative day 1 to day 7
  Pain levels will be assessed daily for 7 days following mandibular third molar surgery using the Visual Analog Scale (VAS), a 10-centimeter scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity. Patients will complete the VAS form daily, and the average score across the 7-day period will be calculated for each participant.
  Unit of Measure: Visual Analog Scale score (0-10)
Total bacterial load on suture materials evaluated by qPCR | Postoperative day 7
  On postoperative day 7, suture materials will be collected from each participant. DNA will be isolated using a commercial extraction kit, and real-time polymerase chain reaction (qPCR) targeting the 16S ribosomal RNA (rRNA) gene will be performed to quantify total bacterial DNA. Results will be expressed as the number of 16S rRNA gene copies per sample.
  Unit of Measure: Copies of 16S rRNA gene per sample
Wound healing status on postoperative day 7 | Postoperative day 7
  The surgical site will be clinically evaluated for wound healing on day 7 after surgery using a standardized Early Wound Healing Index (EHI), which assesses clinical signs such as redness, swelling, bleeding, and epithelialization. The EHI is scored on a scale from 0 to 5, where 0 indicates very poor healing and 5 indicates excellent healing. Higher scores reflect better healing outcomes.
  Unit of Measure: Early Wound Healing Index score (0-5)

SECONDARY OUTCOMES:
Number of analgesic tablets consumed postoperatively | From postoperative day 1 to day 7
  Participants will record the number of analgesic tablets taken each day for 7 days after surgery in a home diary. The total number of tablets consumed will be calculated. Unit of Measure: Number of tablets per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient information will be kept confidential.